CLINICAL TRIAL: NCT03028987
Title: Project 1. The Role of CD4+ Memory Phenotype, Memory, and Effector T-Cells in Vaccination and Infection - Influenza-specific DR1501+ and DR0701+ T-cells
Brief Title: Adaptive Immune Responses and Repertoire in Influenza Vaccination and Infection (SLVP031)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: LAIV was no longer recommended by ACIP
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-31434-2014-2019; 2U19AI057229-11 (NIH)
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-07

CONDITIONS: Influenza
Keywords: Quadrivalent, inactivated influenza vaccine; Quadrivalent, live, attenuated influenza vaccine; Identical twin adults
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LAIV randomized (Other): Volunteers are past participants who have been identified as HLA DR1501+ or DR0701+ by lab assay results. All participants will be randomized within the twin pair to receive either the seasonal quadrivalent live, attenuated influenza vaccine (LAIV4)/ FluMist® or the seasonal quadrivalent inactivated influenza vaccine (IIV4)/ Fluzone® .
  Interventions: Biological: FluMist®
- IIV4 randomized (Other): Volunteers are past participants who have been identified as HLA DR1501+ or DR0701+ by lab assay results. All participants will be randomized within the twin pair to receive either the seasonal quadrivalent live, attenuated influenza vaccine (LAIV4)/ FluMist® or the seasonal quadrivalent inactivated influenza vaccine (IIV4)/ Fluzone®
  Interventions: Biological: Fluzone®

INTERVENTIONS:
Biological: Fluzone® — Fluzone® Quadrivalent (IIV4; inactivated influenza virus vaccine)
  Arms: IIV4 randomized
Biological: FluMist® — FluMist® Intranasal Spray (quadrivalent, live, attenuated influenza vaccine)
  Arms: LAIV randomized

SUMMARY:
The purpose of this study is provide a better understanding of the adaptive immune response to the licensed flu vaccines. The investigators hope the information learned from this study will help identify and describe important factors of influenza immunity especially of or specific proteins associated with the T-cell immune response.

DETAILED DESCRIPTION:
This is a study of up to 20 healthy monozygotic (MZ) twins, 18-49 years old, that are participants from past Stanford-LPCH Vaccine Program trials and who have been identified as human leukocyte antigen (HLA) DR1501+ or DR0701+ by lab assay results. Volunteers will be contacted to assess interest in participating in this study. Both twins in the pair must be willing to participate in the study. All participants will be randomized within the twin pair to receive either the seasonal live, attenuated influenza vaccine (LAIV) or the seasonal quadrivalent inactivated influenza vaccine (IIV4). Immunization will be at Day 0, blood samples for immunogenicity assays will be collected prior to immunization and at Days 7 (6-8) and 28 (24-32).

This study was halted due to the Advisory Committee on Immunization Practices decision not to recommend use of LAIV.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy 18-49 years old identical (MZ) twins identified as DR1501+ or DR0701+ by lab assay results. Both twins in the pair must be willing to participate in the study.
2. Willing to complete the informed consent process
3. Availability for follow-up for the planned duration of the study
4. Acceptable medical history by review of inclusion/exclusion criteria and vital signs.

Exclusion Criteria:

1. Prior off-study vaccination with the current year's seasonal influenza vaccine.
2. Allergy to egg or egg products or to vaccine components including gentamicin, gelatin, arginine or MSG
3. Life-threatening reactions to previous influenza vaccinations
4. Asthma (a contraindication for receipt of LAIV4)
5. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
6. History of immunodeficiency (including HIV infection)
7. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
8. Blood pressure >150 systolic or >95 diastolic at first study visit and the day of vaccination.
9. Hospitalization in the past year for congestive heart failure or emphysema.
10. Chronic Hepatitis B or C.
11. Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible in all groups; inhaled steroid use is not permissible)
12. Participants who care for severely immunosuppressed persons that require a protective environment should not receive LAIV, or should avoid contact with such persons for 7 days after receipt, given the theoretical risk for transmission of the live attenuated vaccine virus to close contacts. [If yes, may be ineligible]
13. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
14. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
15. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
16. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. per day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
17. Has taken an influenza antiviral medication within 48 hours prior to study vaccination [If yes, may not eligible if unable to schedule at an appropriate interval].
18. Receipt of blood or blood products within the past 6 months or planned used during the study.
19. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
20. Receipt of an inactivated vaccine 14 days prior to study enrollment, or planned vaccinations prior to completion of last study visit ( ~ 28 days after study vaccination)
21. Receipt of a live, attenuated vaccine within 60 days prior to enrollment of planned vaccination prior to completion of last study visit (~ 28 days after study vaccination)
22. Need for allergy immunization (that cannot be postponed) during the study period.
23. History of Guillain-Barré syndrome
24. Pregnant or lactating woman
25. Use of investigational agents within 30 days prior to enrollment or planned use during the study.
26. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or planned donation prior to completion of the last visit.
27. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2015-11-18 (Actual); Study Completion 2015-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Dekker, MD, Principal Investigator — Stanford University; Mark Davis, PhD, Principal Investigator — Stanford University; K. Christopher Garcia, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers are past participants who are identical twins and who have been identified as HLA DR1501+ or DR0701+ by lab assay results.
Pre-assignment Details: All participants will be randomized within the twin pair to receive either the seasonal quadrivalent live, attenuated influenza vaccine (LAIV4)/ FluMist® or the seasonal quadrivalent inactivated influenza vaccine (IIV4)/ Fluzone® .
Groups:
- LAIV Randomized: Individual twins in this group received FluMist®: FluMist® Intranasal Spray (quadrivalent, live, attenuated influenza vaccine).
- IIV4 Randomized: Individual twins in this group received Fluzone®: Fluzone® Quadrivalent (IIV4; inactivated influenza virus vaccine).
Period: Overall Study
Arm/Group | LAIV Randomized | IIV4 Randomized
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LAIV Randomized: Individual twins are past participants who have been identified as HLA DR1501+ or DR0701+ by lab assay results. All participants will be randomized within the twin pair to receive either the seasonal quadrivalent live, attenuated influenza vaccine (LAIV4)/ FluMist® or the seasonal quadrivalent inactivated influenza vaccine (IIV4)/ Fluzone® .
  FluMist®: FluMist® Intranasal Spray (quadrivalent, live, attenuated influenza vaccine)
- IIV4 Randomized: Individual twins are past participants who have been identified as HLA DR1501+ or DR0701+ by lab assay results. All participants will be randomized within the twin pair to receive either the seasonal quadrivalent live, attenuated influenza vaccine (LAIV4)/ FluMist® or the seasonal quadrivalent inactivated influenza vaccine (IIV4)/ Fluzone®
  Fluzone®: Fluzone® Quadrivalent (IIV4; inactivated influenza virus vaccine)
- Total: Total of all reporting groups
Arm/Group | LAIV Randomized | IIV4 Randomized | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 46 (9.79) | 46 (9.79) | 46 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Influenza Vaccine
Description: Number of individual twins who received either LAIV or IIV4 as dictated by their group assignment
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV Randomized | IIV4 Randomized
Number analyzed (Participants) | 5 | 5
Participants | 5 | 5

2. Secondary Outcome: Number of Participants With Related Adverse Events
Description: Number of individual twins who experienced related adverse events through the course of the study.
Time Frame: Day 0 to 28 post-immunization
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV Randomized | IIV4 Randomized
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Day 0 to 28 days post-immunization.
Description: Adverse Events will be collected from Day 0 to 28 days post-immunization.
Arm/Group | LAIV Randomized | IIV4 Randomized
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No